CLINICAL TRIAL: NCT02168842
Title: Phase 3 Double-blind Placebo-controlled Parallel Group Study of Isradipine as a Disease Modifying Agent in Subjects With Early Parkinson Disease
Brief Title: Efficacy of Isradipine in Early Parkinson Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Michael J. Fox Foundation for Parkinson's Research (Other); The Parkinson Study Group (Network)
Responsible Party: Principal Investigator, Robert Holloway, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STEADY-PD III; U01NS080818-01A1 (NIH); U01NS080840-01A1 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Parkinson Disease; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Isradipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isradipine (Active Comparator): Oral capsule of up to 5 mg of isradipine taken twice daily for 36 months.
  Interventions: Drug: Isradipine
- Placebo (for Isradipine) (Placebo Comparator): Oral capsule taken twice daily for 36 months.
  Interventions: Drug: Placebo (for Isradipine)

INTERVENTIONS:
Drug: Isradipine — Oral capsules Isradipine IR, up to 10 mg, taken twice daily
  Arms: Isradipine
Drug: Placebo (for Isradipine) — Sugar Pill manufactured to look like Isradipine but has no active ingredients
  Arms: Placebo (for Isradipine)

SUMMARY:
The purpose of the study is to determine whether treatment with isradipine is effective in slowing the progression of Parkinson disease disability.

DETAILED DESCRIPTION:
The study will enroll 336 participants in this multi-center study at approximately 56 sites across the US and Canada. In this study, we are comparing 10 mg of Isradipine to Placebo for treatment of newly diagnosed PD patients. Isradipine has been approved by the Food and Drug Administration (FDA) to treat high blood pressure but is considered investigational in this study, as it has not been approved for use in patients with PD.Isradipine can affect the function of specialized channels that are present in the types of brain cells that are affected in PD patient. These cells are usually responsible for making dopamine, which is depleted in patients with PD. Isradipine may block the damage caused by the flow of certain chemicals through these channels. Laboratory data has showed that Isradipine may prevent the development of Parkinson-like symptoms in animal studies. Isradipine has been evaluated in some patients with PD. The first study with isradipine controlled release (CR) in patients with early PD and normal blood pressure found that the drug was reasonably well tolerated and safe. The controlled release formulation of isradipine is not available for use and therefore this study is using the immediate release formulation. Eligible participants will be followed for up to 36 months and will be expected to complete 12 in-person visits and 4 telephone visits. The study visits will include clinical assessment of motor, neuropsychiatric and cognitive testing as well as collection of blood and urine samples. Study drug will taken twice daily, in the morning and in the evening with or without food. Prior to taking study drug, study participants will be required to take their blood pressure with a home blood pressure device provided to them for use in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with early idiopathic PD (presence of at least two out of three cardinal manifestations of PD). If tremor is not present, subjects must have unilateral onset and persistent asymmetry of the symptoms
* Age equal or greater than 30 years at the time of diagnosis of PD
* Hoehn and Yahr stage less than or equal to 2
* Diagnosis of PD less than 3 years.
* Currently NOT receiving dopaminergic therapy (levodopa, dopamine agonist or MAO-B inhibitors) and NOT projected to require PD symptomatic therapy for at least 3 months from the baseline visit
* Use of amantadine and/or anticholinergics will be allowed provided that the dose is stable for 8 weeks prior to the baseline visit
* If subject is taking any central nervous system acting medications (e.g., benzodiazepines, antidepressants, hypnotics) regimen must be stable for 30 days prior to the baseline visit
* Women of childbearing potential may enroll but must use a reliable measure of contraception and have a negative serum pregnancy test at the screening visit

Exclusion Criteria:

* Subjects with a diagnosis of an atypical Parkinsonism
* Subjects unwilling or unable to give informed consent
* Exposure to dopaminergic PD therapy within 60 days prior to baseline visit or for consecutive 3 months or more at any point in the past
* History of clinically significant orthostatic hypotension or presence of orthostatic hypotension at the screening or baseline visit defined as greater than or equal to 20 mmHg change in systolic BP and greater than or equal to 10 mmHg change in diastolic BP from sitting position to standing after 2 minutes, or baseline sitting BP less than 90/60
* History of congestive heart failure
* Clinically significant bradycardia
* Presence of 2nd or 3rd degree atrioventricular block or other significant ECG abnormalities that in the investigator's opinion would compromise participation in study
* Clinically significant abnormalities in the Screening Visit laboratory studies or ECG
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* Prior exposure to isradipine or other dihydropyridine calcium channel blockers within 6 months of the baseline visit
* Subjects on greater than 2 concomitant antihypertensive medications. If a history of hypertension, then a maximum of 2 other antihypertensive agents will be allowed provided that the dosages of concomitant anti HTN therapy can be reduced/adjusted during the study based on the BP readings in consultation with the subject's primary care provider or cardiologist. Use of any concomitant calcium channel blockers will not be allowed from the baseline visit and for the duration of the study
* Use of grapefruit juice, ginkgo biloba, St. John's wort or ginseng will be prohibited starting from the screening visit and for the duration of the study (as they interfere with the metabolism of isradipine)
* Use of clarithromycin, telithromycin and erythromycin will be prohibited starting from the screening visit and for the duration of the study as the combination of clarithromycin, telithromycin or erythromycin and calcium channel blockers has been reported to be associated with increased risk of kidney and heart injury
* Presence of cognitive dysfunction defined by a Montreal Cognitive assessment (MoCA) score of less than 26 at screening
* Subjects with clinically significant depression as determined by a Beck Depression Inventory II (BDI) score greater than 15 at the screening visit
* History of exposure to typical or atypical antipsychotics or other dopamine blocking agents within 6 months prior to the baseline visit
* History of use of an investigational drug within 30 days prior to the screening visit
* History of brain surgery for PD
* Allergy/sensitivity to isradipine or its matching placebo or their formulations
* Pregnant or lactating woman

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, MD, Principal Investigator — Northwestern University; Robert Holloway, MD MPH, Principal Investigator — University of Rochester
Locations (54):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Sun Health Research Institute, Sun City, Arizona
  - The Parkinsons & Movement Disorder Institute, Fountain Valley, California
  - University of California, Irvine, California
  - University of California San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Institute of Neurodegenerative Disorders, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Pacific Health Research & Education Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - LSU Health Science Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Atlantic Neuroscience Institute, Summit, New Jersey
  - Albany Medical College, Albany, New York
  - Health Quest Kingston, Kingston, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Ottawa Hospital Civic Site, Ottawa, Ontario
  - The Centre for Addiction and Mental Health, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - Centre Hospitalier Affilie, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Di Luca DG, Macklin EA, Hodgeman K, Lopez G, Pothier L, Callahan KF, Lowell J, Chan J, Videnovic A, Lungu C, Lang AE, Litvan I, Schwarzschild MA, Simuni T. Enrollment of Participants From Marginalized Racial and Ethnic Groups: A Comparative Assessment of the STEADY-PD III and SURE-PD3 Trials. Neurol Clin Pract. 2023 Feb;13(1):e200113. doi: 10.1212/CPJ.0000000000200113. Epub 2023 Jan 18. PMID 36865634
- [Derived] Venuto CS, Yang L, Javidnia M, Oakes D, James Surmeier D, Simuni T. Isradipine plasma pharmacokinetics and exposure-response in early Parkinson's disease. Ann Clin Transl Neurol. 2021 Mar;8(3):603-612. doi: 10.1002/acn3.51300. Epub 2021 Jan 18. PMID 33460320
- [Derived] Parkinson Study Group STEADY-PD III Investigators. Isradipine Versus Placebo in Early Parkinson Disease: A Randomized Trial. Ann Intern Med. 2020 May 5;172(9):591-598. doi: 10.7326/M19-2534. Epub 2020 Mar 31. PMID 32227247
- [Derived] McFarthing K, Simuni T. Clinical Trial Highlights: Phase III Study in Spotlight. J Parkinsons Dis. 2019;9(1):3-4. doi: 10.3233/JPD-190002. No abstract available. PMID 30741695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 57 Parkinson Study Group sites in North America from November 2014 through November 2015.
Pre-assignment Details: 413 patients were assessed for eligibility. 12 patients declined to participate and 65 patients were excluded (9 exclusionary medications, 2 other medical psychiatric or surgical, 5 disease too advanced, 6 diagnosis uncertain, 23 didn't meet other inclusion criteria, 20 other). 336 patients were enrolled and underwent randomization
Groups:
- Isradipine: Receive Isradipine 5 mg twice daily for 36 months. Isradipine: oral immediate-release capsule of Isradipine 10 mg per day.
- Placebo (for Isradipine): Receive placebo twice daily for 36 months. Placebo: Sugar Pill manufactured to look like Isradipine but has no active ingredients
Period: Overall Study
Arm/Group | Isradipine | Placebo (for Isradipine)
Started | 170 | 166
Completed | 162 | 158
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 2 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isradipine | Placebo (for Isradipine) | Total
Number analyzed (Participants) | 170 | 166 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.11 (8.73) | 61.61 (9.34) | 61.86 (9.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 58 | 106
  Male | 122 | 108 | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 166 | 160 | 326
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 7 | 10
  White | 159 | 149 | 308
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants] — Enrolled patients were from 54 Parkinson Study Group sites in North America. 7 locate in Canada and 47 locate in United States.
  participants
    United States | 154 | 149 | 303
    Canada | 16 | 17 | 33
Disease Duration [Mean (Standard Deviation); unit: months] — Months from diagnosis.
  months | 9.89 (8.13) | 10.56 (9.35) | 10.22 (8.75)
Family History of PD [Count of Participants; unit: Participants] — First degree relatives only
  Participants | 30 | 35 | 65
Handedness [Count of Participants; unit: Participants]
  Right | 147 | 142 | 289
  Left | 20 | 19 | 39
  Mixed | 3 | 5 | 8
On Symptomatic Therapy (Amantadine) [Count of Participants; unit: Participants] | 15 | 11 | 26
On Symptomatic Therapy (Anticholinergics) [Count of Participants; unit: Participants] | 3 | 2 | 5
UPDRS Total Score [Mean (Standard Deviation); unit: units on a scale] — Baseline total Unified Parkinson Disease Rating Scale (UPDRS) score ranges from 0 to 52. Larger value stands for more disability from PD. Population: One participant had missing baseline UPDRS
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 23.66 (8.64) | 22.58 (8.53) | 23.13 (8.59)
Mental Scale [Mean (Standard Deviation); unit: units on a scale] — Baseline UPDRS Mental (UPDRS Part I: Mentation, Behavior, and Mood) score ranges from 0 to 7. Larger value stands for more disability from PD. Population: One participant had missing baseline UPDRS
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 0.61 (0.87) | 0.81 (1.21) | 0.71 (1.05)
ADL Scale [Mean (Standard Deviation); unit: units on a scale] — Baseline UPDRS ADL (Part II) score ranges from 0 to 16. Larger value stands for more disability from PD. UPDRS Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food. Population: One participant had missing baseline UPDRS
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 4.96 (2.88) | 5.45 (3.26) | 5.2 (3.08)
Motor Scale [Mean (Standard Deviation); unit: units on a scale] — Baseline UPDRS Motor (Part III) score ranges from 0 to 42. Larger value stands for more disability from PD. UPDRS part III: clinician-scored monitored motor evaluation Population: One participant had missing baseline UPDRS
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 18.08 (7.3) | 16.32 (6.53) | 17.21 (6.97)
UPSDRS PIGD Score [Mean (Standard Deviation); unit: units on a scale] — Baseline UPDRS PIGD score ranges from 0 to 1. Larger value stands for more disability from PD. Population: One participant had missing baseline UPDRS PIGD Score
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 0.17 (0.19) | 0.17 (0.17) | 0.17 (0.18)
UPDRS Tremor Score [Mean (Standard Deviation); unit: units on a scale] — Baseline UPDRS Tremor score ranges from 0 to 1.63. Larger value stands for more disability from PD. Population: One participant had missing baseline UPDRS Tremor Score
  units on a scale
    number analyzed (Participants) | 170 | 165 | 335
    (all) | 0.51 (0.32) | 0.50 (0.29) | 0.51 (0.3)
H/Y Stage [Mean (Standard Deviation); unit: units on a scale] — Hoehn and Yahr staging of severity of Parkinson's disease. Baseline H/Y stage ranges from 1 to 3. Larger value stands for more disability from PD.
  units on a scale | 1.72 (0.46) | 1.6 (0.5) | 1.66 (0.48)
SE/ADL [Mean (Standard Deviation); unit: units on a scale] — Schwab and England ADL scale. Baseline SE/ADL ranges from 40 to 100. Smaller value stands for more disability from PD.
  units on a scale | 94.44 (5.23) | 94.04 (6.8) | 94.24 (6.05)
Modified Rankin Score [Mean (Standard Deviation); unit: units on a scale] — The modified Rankin Scale (mRS) measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Baseline Modified Rankin score ranges from 0 to 2. Larger value stands for more disability from PD.
  units on a scale | 1.09 (0.31) | 1.09 (0.33) | 1.09 (0.32)
MoCA Score [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MoCA) is one-page 30-point test to detect cognitive impairment. Baseline MoCA score ranges from 23 to 30. Higher scores indicate better cognition.
  units on a scale | 28.14 (1.41) | 28.04 (1.29) | 28.09 (1.35)
BDI Total Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Beck Depression Inventory (BDI) score ranges from 0 to 23. Higher scores indicate greater symptom severity.
  units on a scale | 4.09 (3.71) | 4.8 (4.29) | 4.44 (4.02)
PDQ39 Total Score [Mean (Standard Deviation); unit: units on a scale] — Parkinson's Disease Questionnaire-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the past month. Baseline PDQ 39 score ranges from 0 to 52. Lower score shows better quality of life.
  units on a scale | 7.13 (6.15) | 9.08 (8.52) | 8.10 (7.47)
Systolic BP, Seated [Mean (Standard Deviation); unit: mmHg] | 128.12 (17.17) | 127.69 (14.6) | 127.91 (15.93)
Diastolic BP, Seated [Mean (Standard Deviation); unit: mmHg] | 76.55 (9.72) | 77.83 (8.52) | 77.18 (9.16)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in Total Unified Parkinson Disease Rating Scale (UPDRS) Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the total (Part I-III) UPDRS score in the active treatment arm versus placebo between the baseline and 36 month visit. The change of UPDRS ranges from -30 to 80, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 2.99 [0.95 to 5.03] | 3.26 [1.25 to 5.26]

2. Primary Outcome: Adjusted Mean Change in Adjusted UPDRS Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the adjusted UPDRS Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change of adjusted UPDRS ranges from -100 to 150, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 13.49 [11.32 to 15.66] | 13.85 [11.72 to 15.98]

3. Secondary Outcome: Adjusted Mean Change in LED
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the LED(levodopa equivalent dose) in the active treatment arm versus placebo between the baseline and 36 month visit. The change of LED ranges from -100 to 3000, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline LED measurement. So LED had 1 more observation than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mg | 389 [337 to 441] | 375 [325 to 426]

4. Secondary Outcome: Adjusted Mean Change in LED Cumulative
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the LED(levodopa equivalent dose) cumulative in the active treatment arm versus placebo between the baseline and 36 month visit. The change of LED cumulative ranges from 0 to 1200000, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline LED Cumulative measurement. So LED Cumulative had 1 more observation than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mg | 676 [588 to 765] | 697 [611 to 784]

5. Secondary Outcome: Adjusted Mean Change in UPDRS Part IV
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the UPDRS Part IV in the active treatment arm versus placebo between the baseline and 36 month visit. The change in UPDRS Part IV ranges from -10 to 10, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. 46 patients had missing measures at the visit of 36 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 134 | 140
score on a scale | 1.18 [0.9 to 1.46] | 1.07 [0.8 to 1.33]

6. Secondary Outcome: Adjusted Mean Change in MDS-UPDRS nmEDL
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the MDS-UPDRS nmEDL(Non-Motor Experiences of Daily Living) in the active treatment arm versus placebo between the baseline and 36 month visit. The change in MDS-UPDRS nmEDL ranges from -6 to 10, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 1.93 [1.28 to 2.59] | 1.76 [1.13 to 2.4]

7. Secondary Outcome: Adjusted Mean Change in MDS-UPDRS mEDL
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the MDS-UPDRS mEDL(Motor Experiences of Daily Living) in the active treatment arm versus placebo between the baseline and 36 month visit. The change in MDS-UPDRS mEDL ranges from -8 to 35, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 2.32 [1.52 to 3.12] | 2.57 [1.78 to 3.35]

8. Secondary Outcome: Adjusted Mean Change in UPDRS Score to 1 Year
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the MDS-UPDRS nmEDL(Non-Motor Experiences of Daily Living) in the active treatment arm versus placebo between the baseline and 12 month visit. The change of UPDRS ranges from -22 to 23, larger value shows more disability from PD.
Time Frame: Baseline to 12 months of treatment
Population: Intention-to-treat (ITT) population. There were 169 patients in Isradipine group and 165 in placebo group who reached 1-year visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 169 | 165
score on a scale | 4.65 [3.59 to 5.70] | 5.3 [4.25 to 6.35]

9. Secondary Outcome: Adjusted Mean Change in UPDRS Part II
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the UPDRS Part II (ADL Function) in the active treatment arm versus placebo between the baseline and 36 month visit. The change in UPDRS Part II ranges from -12 to 19, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 2.3 [1.63 to 3.97] | 2.5 [1.83 to 3.16]

10. Secondary Outcome: Adjusted Mean Change in UPDRS Part III OFF
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the UPDRS Part III OFF rating in the active treatment arm versus placebo between the baseline and 36 month visit. The change in UPDRS Part III OFF ranges from -30 to 100, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. 58 patients had missing measures at the visit of 36 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 129 | 133
score on a scale | 4.60 [3.05 to 6.14] | 4.50 [3.02 to 5.98]

11. Secondary Outcome: Adjusted Mean Change in SE/ADL
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the SE/ADL in the active treatment arm versus placebo between the baseline and 36 month visit. The change of UPDRS ranges from -70 to 20, larger value shows improvement of PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline SE/ADL measurement. So SE/ADL had 1 more observation than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
units on a scale | -4.14 [-5.30 to -2.98] | -4.41 [-5.54 to -3.27]

12. Secondary Outcome: Adjusted Mean Change in Modified Rankin Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Modified Rankin Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in Modified Rankin Score ranges from -1 to 3, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline measurement for primary efficacy while had finished baseline Modified Rankin Score. So Modified Rankin Score had 1 more observation than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
units on a scale | 0.18 [0.07 to 0.28] | 0.29 [0.18 to 0.39]

13. Secondary Outcome: Adjusted Mean Change in MoCA Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the MoCA Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in MoCA Score ranges from -10 to 6, larger value shows improvement of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline MoCA Score. So MoCA Score had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
units on a scale | -0.04 [-0.36 to 0.28] | -0.07 [-0.39 to 0.25]

14. Secondary Outcome: Adjusted Mean Change in PDQ39 Total Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the PDQ39 Total Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in PDQ39 Total Score ranges from -16 to 44, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. 7 patients had missing PDQ39 scores at the visit of 36 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 158 | 155
units on a scale | 2.80 [1.42 to 4.18] | 3.42 [2.07 to 4.77]

15. Secondary Outcome: Adjusted Mean Change in Ambulatory Capacity
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Ambulatory Capacity in the active treatment arm versus placebo between the baseline and 36 month visit. The change in Ambulatory Capacity ranges from -4 to 12, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
score on a scale | 0.59 [0.34 to 0.85] | 0.50 [0.25 to 0.75]

16. Secondary Outcome: Adjusted Mean Change in BDI Total Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the BDI Total Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in BDI Total Score ranges from -9 to 22, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant in Placebo group had missing baseline UPDRS sections while had finished baseline BDI Score. And one participant in Isradipine group had missing BDI score at the visit of 36 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 161 | 159
units on a scale | 0.77 [0.05 to 1.49] | 1.34 [0.63 to 2.04]

17. Secondary Outcome: Risk of Need for Antiparkinsonian Therapy
Description: Number of participants with need for Antiparkinsonian Therapy.
Time Frame: Baseline to 36 months of treatment
Population: Include all 336 patients that were randomized, no matter whether or not completed the study.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 170 | 166
participants | 145 [134 to 153] | 147 [138 to 154]
Statistical Analysis 1: Comparison: Isradipine vs Placebo (for Isradipine); Test type: Equivalence — Comparison of the risk of need for antiparkinsonian therapy in Isradipine group to the risk in placebo group; p = 0.073, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.61 to 1.03]

18. Secondary Outcome: Risk of Need for Dyskinesia
Description: Number of participants with need for Dyskinesia Therapy.
Time Frame: Baseline to 36 months of treatment
Population: Include all 336 patients that were randomized, no matter whether or not completed the study.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 170 | 166
participants | 24 [17 to 34] | 19 [12 to 28]
Statistical Analysis 1: Comparison: Isradipine vs Placebo (for Isradipine); Test type: Equivalence — Comparison the risk of need for dyskinesia in Isradipine group to the risk in a placebo group; p = 0.21, Log Rank; Hazard Ratio (HR) = 1.53, 95% CI 2-sided [0.78 to 3.01]

19. Secondary Outcome: Risk of Need for Fluctuations
Description: Number of participants with need for Fluctuations Therapy.
Time Frame: Baseline to 36 months of treatment
Population: Include all 336 patients that were randomized, no matter whether or not completed the study.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 170 | 166
participants | 57 [46 to 70] | 64 [51 to 76]
Statistical Analysis 1: Comparison: Isradipine vs Placebo (for Isradipine); Test type: Equivalence — Comparison of the risk of need for antiparkinsonian therapy in Isradipine group to the risk in placebo group; p = 0.35, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.56 to 1.22]

20. Other Pre Specified Outcome: Adjusted Mean Change in UPDRS PIGD Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the UPDRS PIGD Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in UPDRS PIGD Score ranges from -1 to 3, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
units on a scale | 0.12 [0.07 to 0.17] | 0.10 [0.05 to 0.15]

21. Other Pre Specified Outcome: Adjusted Mean Change in UPDRS Tremor Score
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the UPDRS Tremor Score in the active treatment arm versus placebo between the baseline and 36 month visit. The change in UPDRS Tremor Score ranges from -1 to 2, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 158
units on a scale | 0.00 [-0.05 to 0.05] | 0.01 [-0.03 to 0.06]

22. Other Pre Specified Outcome: Adjusted Mean Change in H/Y Stage
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the H/Y Stage in the active treatment arm versus placebo between the baseline and 36 month visit. The change in H/Y Stage ranges from -1 to 3, larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline H/Y Stage. So H/Y Stage had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
units on a scale | 0.15 [0.09 to 0.22] | 0.21 [0.15 to 0.28]

23. Other Pre Specified Outcome: Adjusted Mean Change in Levodopa
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Levodopa in the active treatment arm versus placebo between the baseline and 36 month visit. The change of LED ranges from -200 to 2000, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline Levodopa. So Levodopa had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mg | 307 [257 to 356] | 307 [259 to 355]

24. Other Pre Specified Outcome: Adjusted Mean Change in Levodopa Cumulative
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Levodopa Cumulative in the active treatment arm versus placebo between the baseline and 36 month visit. The change of Levodopa cumulative ranges from 0 to 800000, larger value shows more disability from PD.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline Levodopa Cumulative. So Levodopa Cumulative had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mg | 471 [388 to 555] | 508 [426 to 590]

25. Other Pre Specified Outcome: Adjusted Mean Change in Systolic BP, Seated
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Systolic BP, Seated in the active treatment arm versus placebo between the baseline and 36 month visit. The change in Systolic BP, Seated ranges from -65 to 50. larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline Systolic BP, Seated. So Systolic BP had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mmHg | -6.11 [-8.28 to -3.95] | 1.03 [-1.10 to 3.15]

26. Other Pre Specified Outcome: Adjusted Mean Change in Diastolic BP, Seated
Description: Efficacy of isradipine to slow progression of Parkinson disease disability to be determined by the change in the Diastolic BP, Seated in the active treatment arm versus placebo between the baseline and 36 month visit. The change in Diastolic BP, Seated ranges from -35 to 25. larger value shows worsening of conditions.
Time Frame: Baseline to 36 months of treatment
Population: Intention-to-treat (ITT) population. One participant had missing baseline UPDRS sections while had finished baseline Diastolic BP, Seated. So Diastolic BP had 1 observation more than primary outcomes.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Isradipine | Placebo (for Isradipine)
Number analyzed (Participants) | 162 | 159
mmHg | -4.64 [-5.93 to -3.36] | -0.71 [-1.96 to 0.55]

ADVERSE EVENTS:
Time Frame: Baseline to 36 months of treatment
Arm/Group | Isradipine | Placebo (for Isradipine)
All-Cause Mortality (participants affected / at risk) | 2/170 | 1/166
Serious Adverse Events (participants affected / at risk) | 26/170 | 27/166
Other Adverse Events (participants affected / at risk) | 163/170 | 154/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isradipine (N=170) | Placebo (for Isradipine) (N=166)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0)
STRESS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 2 (2) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1)
APPENDICEAL MUCOCOELE (Gastrointestinal disorders) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHOROID MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
PANCREATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SPINA BIFIDA (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
THROAT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isradipine (N=170) | Placebo (for Isradipine) (N=166)
DIZZINESS (Nervous system disorders) | 42 (55) | 26 (30)
NAUSEA (Gastrointestinal disorders) | 26 (29) | 32 (38)
HEADACHE (Nervous system disorders) | 28 (40) | 17 (19)
OEDEMA (General disorders) | 31 (41) | 9 (11)
NASOPHARYNGITIS (Infections and infestations) | 23 (26) | 22 (23)
FATIGUE (General disorders) | 23 (28) | 20 (21)
CONSTIPATION (Gastrointestinal disorders) | 23 (24) | 21 (22)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 (19) | 20 (26)
INSOMNIA (Psychiatric disorders) | 19 (22) | 19 (20)
ANXIETY (Psychiatric disorders) | 20 (22) | 13 (16)
DEPRESSION (Psychiatric disorders) | 20 (22) | 13 (14)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 17 (20) | 15 (16)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (13) | 11 (20)
FALL (Injury, poisoning and procedural complications) | 7 (10) | 15 (20)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 12 (14) | 15 (15)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 (12) | 13 (15)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (14) | 9 (11)
SINUSITIS (Infections and infestations) | 7 (8) | 13 (17)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 9 (11)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 12 (13) | 7 (8)
SOMNOLENCE (Nervous system disorders) | 10 (11) | 8 (9)
HYPOAESTHESIA (Nervous system disorders) | 8 (11) | 6 (8)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (9)
SLEEP DISORDER (Psychiatric disorders) | 9 (9) | 8 (8)
BRONCHITIS (Infections and infestations) | 5 (5) | 11 (12)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (6) | 9 (11)
HYPERTENSION (Vascular disorders) | 8 (8) | 8 (8)
DIARRHOEA (Gastrointestinal disorders) | 7 (11) | 5 (5)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 5 (8)
CATARACT (Eye disorders) | 4 (6) | 7 (9)
DYSPHAGIA (Gastrointestinal disorders) | 7 (9) | 4 (6)
POLLAKIURIA (Renal and urinary disorders) | 7 (7) | 7 (7)
TREMOR (Nervous system disorders) | 5 (5) | 9 (9)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 7 (8) | 6 (6)
RAPID EYE MOVEMENTS SLEEP ABNORMAL (Psychiatric disorders) | 7 (8) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 8 (9)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
DYSTONIA (Nervous system disorders) | 8 (8) | 4 (5)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5)
NEPHROLITHIASIS (Renal and urinary disorders) | 5 (9) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (6)
CHEST PAIN (General disorders) | 6 (7) | 5 (5)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 5 (6) | 6 (6)
INFLUENZA (Infections and infestations) | 3 (3) | 8 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (7) | 4 (4)
MICTURITION URGENCY (Renal and urinary disorders) | 7 (8) | 3 (3)
DIVERTICULITIS (Infections and infestations) | 5 (6) | 1 (5)
LACERATION (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
HYPOTENSION (Vascular disorders) | 4 (4) | 5 (6)
PARAESTHESIA (Nervous system disorders) | 5 (5) | 4 (5)
VISION BLURRED (Eye disorders) | 7 (8) | 2 (2)
ABNORMAL LOSS OF WEIGHT (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 6 (6) | 3 (3)
BLOOD CREATININE INCREASED (Investigations) | 7 (7) | 2 (2)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 7 (7) | 2 (2)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
SCIATICA (Nervous system disorders) | 4 (6) | 3 (3)
VERTIGO (Ear and labyrinth disorders) | 2 (3) | 5 (6)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 5 (5) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 4 (4)
INGUINAL HERNIA (Gastrointestinal disorders) | 4 (4) | 4 (4)
PALPITATIONS (Cardiac disorders) | 6 (6) | 2 (2)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 3 (3) | 5 (5)
FLUSHING (Vascular disorders) | 7 (8) | 0 (0)
BRADYKINESIA (Nervous system disorders) | 3 (3) | 4 (4)
DRY EYE (Eye disorders) | 3 (3) | 4 (4)
HALLUCINATION (Psychiatric disorders) | 1 (1) | 6 (6)
PAIN (General disorders) | 5 (5) | 2 (2)
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 5 (5)
VOMITING (Gastrointestinal disorders) | 3 (3) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 3 (3)
HOT FLUSH (Vascular disorders) | 5 (6) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2 (3) | 4 (4)
TACHYCARDIA (Cardiac disorders) | 4 (5) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 (3) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
AMNESIA (Nervous system disorders) | 3 (3) | 3 (3)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
SYNCOPE (Nervous system disorders) | 4 (4) | 2 (2)
TOOTH ABSCESS (Infections and infestations) | 4 (4) | 2 (2)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
IRRITABILITY (General disorders) | 2 (3) | 3 (3)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (3)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 3 (4) | 1 (2)
ABNORMAL DREAMS (Psychiatric disorders) | 3 (3) | 2 (2)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 3 (3) | 2 (2)
COGNITIVE DISORDER (Nervous system disorders) | 2 (2) | 3 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 5 (5) | 0 (0)
EYE INFECTION (Infections and infestations) | 3 (3) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 3 (3)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 3 (3) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 2 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
PNEUMONIA (Infections and infestations) | 1 (1) | 3 (4)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
ASTHENIA (General disorders) | 2 (2) | 2 (2)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 1 (1)
EAR DISCOMFORT (Ear and labyrinth disorders) | 3 (3) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 4 (4)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 3 (3)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 3 (3) | 1 (1)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 4 (4)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT02168842/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT02168842/SAP_001.pdf